CLINICAL TRIAL: NCT04319393
Title: Testing the Effectiveness of Cognitive Behavioral Therapy in Relieving Nurses' Ageism Toward Older Adults
Brief Title: Cognitive Behavioral Therapy and Ageism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20180217
Record Dates: First submitted 2020-03-19; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Ageism
Keywords: Cognitive Behavioral Therapy; Older Adults; Nurses; Death anxiety; Randomized Clinical Trials
MeSH Terms: conditions — Ageism; Necrophobia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT Nurses (Experimental): Interventional group
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Consultation Nurses (No Intervention): Control Group

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The CBT intervention was carried out through six two-hour sessions over a month. The intervention group was divided into three subgroups of 18 to 19 nurses each. It was required for each subgroup to attend two CBT sessions to complete the intervention.
  The CB therapist followed the same structure in the delivery of each CBT session. The CBT session was delivered in five modules: generating objectives and outcomes, enhancing self-esteem and interpersonal relationships, changing beliefs regarding symbolic mortality, and changing attitudes regarding death anxiety. The first session began with highlighting the objectives of the CBT. Then, a detailed presentation of the intervention modules was provided to the nurses with integration of CBT exercises, including cognitive restructuring, graded exposure, mindfulness meditation, interpersonal skills training, and activity scheduling
  Arms: CBT Nurses

SUMMARY:
Background: Healthcare settings must be a patient-friendly environment for the investigator's older adults who are in an imperative need for compassionate healthcare when approaching their later life. However, older adults until this moment are experiencing age discriminative acts by nurses who are supposed to act in favor of their patients. Ageism is not always a result of either negative attitudes or misconceptions toward older adults, but to the innate fear of death where nurses perceive older adults as a powerful reminder of death. Although cognitive-behavioral therapy (CBT) is well known for targeting psychological distresses, to date, no research has investigated its effectiveness in relieving nurses' death anxiety and ageism. This study examined the effectiveness of CBT to relieve nurses' death anxiety and ageism toward older adults.

Methods: A randomized controlled trial was conducted during August 2019 in the university hospital. A total of 110 nurses selected through proportional stratified sampling and randomly assigned to the experimental and control groups. The intervention consisted of six two-hour training sessions delivered in five modules with the integration of different CBT exercises. The effect of CBT was assessed on measures of a series of validated questionnaires of study variables before and after the training sessions.

DETAILED DESCRIPTION:
Procedure After getting the IRB approval and completing the informed consent procedure, the researchers met with the administrator of the hospital to (1) discuss the inclusion criteria and obtain a list of eligible participants, (2) discuss the workflow of the study procedure, and (3) agree on the time/date of site visits to collect the data and run the CBT sessions based on the convenience of nurses and their work schedule. After having a list of all eligible nurses recorded in an excel sheet, the researcher randomly assigned the nurses into control and intervention groups using Excel's RAND function. After randomization was performed, the researchers distributed the pretest questionnaires to the nurses in both groups and asked them to drop the completed questionnaires in the designated box next to the front desk of their work department. Three days later the researchers collected the questionnaires.

Intervention The CBT intervention was carried out through six two-hour sessions over a month. The intervention group was divided into three subgroups of 18 to 19 nurses each. It was required for each subgroup to attend two CBT sessions to complete the intervention. The main objective of the CBT was to improve nurses' senses of self-esteem, interpersonal relationship, and symbolic immortality. The CBT was guided by the five-factor model, which extensively used within the context of CBT (Bagby, Gralnick, Al-Dajani, & Uliaszek, 2016). A detailed description of the model was discussed in previous recent studies (Bagby et al., 2016; Hawley et al., 2017). The model explains the interactions between beliefs, attitudes, emotions, and behaviors. The intervention emphasized on how nurses can reinforce and enhance their anxiety buffering system by an improved understanding of how unconscious realization of eventual mortality affects explicit attitudes. Throughout the intervention, nurses were trained about the five-factor model and therapeutic beliefs, emotions, attitudes, and behaviors pertinent to death anxiety. The differences between therapeutic and nontherapeutic coping strategies of death anxiety were identified and discussed with nurses in the intervention group.

The CB therapist followed the same structure in the delivery of each CBT session. The CBT session was delivered in five modules: generating objectives and outcomes, enhancing self-esteem and interpersonal relationships, changing beliefs regarding symbolic mortality, and changing attitudes regarding death anxiety. The CBT was tailored to meet the training needs of nurses based on the analysis of pretest questionnaire scores. The first session began with highlighting the objectives of the CBT. Then, a detailed presentation of the intervention modules was provided to the nurses with the integration of CBT exercises, including cognitive restructuring, graded exposure, mindfulness meditation, interpersonal skills training, and activity scheduling.

. At the end of the first session, the nurses were assigned to solve some homework questions relevant to the CBT exercises. The second session began with a brainstorming of the CBT training assignments from the first session. Then thoughts and understandings of training assignments and reflection on life stories or real experiences of alternative therapeutic behaviors were discussed. The CBT therapist was an experienced certified psychologist with a Ph.D. degree in Applied Psychology.

The nurses in the control group were divided into the same number of subgroups as the CBT nurses and trained by an experienced gerontological nurse who provided two consultations of 120 minutes for each subgroup. The main objective of the consultations was to instruct the nurses on how to deal with or care for older adults with respect and dignity as well as eliminate any ageist attitudes that they might have. The control group did not receive active advice or referrals to a psychologist or CBT therapist. During the consultations, the nurses received written and verbal information about the atypical presentation of illnesses and the most common misconceptions related to aging. The nurses in the control group had the opportunity to discuss and reflect on their own experiences in caring for older adults and other geriatric care-related issues. The consultations were nurse-centered, goal-oriented, and guided by nurses' questions. On the last day of the training for each group (intervention and control), the nurses were asked to fill out the posttest questionnaires and return them to the researchers.

Measures Outcome variables were measured twice; pre and posttest. The primary outcomes in the current were death anxiety and ageism, while the secondary outcomes self-esteem, interpersonal relationship, and symbolic immortality.

Primary Outcome Measures Death anxiety. Death anxiety was measured using The revised Collett-Lester Fear of Death Scale (CL-FODS) (Lester & Abdel-Khalek, 2003). The CL-FODS is a 28-item scale measure death anxiety about four main aspects of death and dying, including: " your own death,"; "your own dying"; " the death of others,"; and " the dying of other". Each subscale has seven items answered on a 3-point intensity scale (ranged from 1= "no" to 5= "very"). The CL-FODS had very satisfactory reliability scores ranged from .88 to .93, and good internal consistency scores ranged from .74 to .90 in the original study. In the current study, the internal consistency reliability was satisfactory (Cronbach's alpha= 0.79) Ageism. The Fraboni Scale of Ageism (FSA) (Fraboni et al., 1990) was used to measure nurses' ageist attitudes toward older adults. The FSA is a 29-item scale measuring the attitudinal and affective aspects of ageism. The FSA has three positive items (e.g., "Old people can be very creative"), which were reverse coded before calculating the total score. Each item of the FSA has four possible responses, including: "1= strongly disagree,"; "2= disagree,"; " 3=agree,"; and " 4= strongly agree". The possible range of the total score of the FSA is from 29 to 116. Higher scores indicate greater levels of ageist attitudes. The internal consistency reliability of the FSA in this study was high (Cronbach's alpha = 0.89), which is very close to the original research (0.86) (Fraboni et al., 1990) Secondary Outcome Measures Self-esteem. Nurses' self-esteem was measured using the Rosenberg Self-Esteem Scale (RSES) (Rosenberg, 2015). The RSES has five positive (e.g., "I take a positive attitude toward myself") and five negatives (e.g., "I feel I do not have much to be proud of") items. The nurses responded to these items using a 4-point Likert scale ranging from 1= "strongly disagree" to 4= "strongly agree." The total score of the RSES was calculated after reverse coding of the negative items yielding a range from 10 to 40, with higher scores indicating greater levels of self-esteem. The Cronbach's alpha reliability of the RSES in this study was high (0.91) Interpersonal relationship. Nurses' interpersonal relationships were measured using the Interpersonal Reactivity Index (IRI) (Davis, 1980). The IRS has four subscales consisting of five positive and two negative items each. The subscales include perspective-taking, fantasy, empathic concern, and personal distress. The nurses responded to the 28 items of IRS with five responses ranging from 0=" Does not describe me well" to 4= "describes me very well." The total score of the IRS was calculated after reverse coding the negative items, yielding a range from 0 to 112. The Cronbach's alpha reliability of the IRI in this study was very good (0.81) Symbolic immortality. Symbolic immortality was measured using the Sense of Symbolic Immortality Scale (SSIS) (Drolet, 2007). The SSIS contains 11 negatives (e.g., nothing interesting happens in my life) and positive (e.g., I feel that I am doing what I want in life) items about areas of life showing the desire for symbolic immortality. The nurses responded to these items using a Likert scale of five choices ranging from 1 = "strongly disagree," to 5 = "strongly agree." The total score of the SSIS was calculated after reverse coding the negative items, yielding a range from 26 to130. Higher scores indicate a greater sense of symbolic immortality. The SSIS had good internal consistency in this study (Cronbach alpha = 0.86).

Other Measures Demographic questionnaire. The demographic data of nurses such as age, gender, level of education, years of clinical experience, marital status, and the number of older adults living in their households were collected by asking the nurses to fill out the demographic questionnaire.

Data Analysis IBM SPSS Statistics for Windows, Version 25.0. (Armonk, NY: IBM Corp) was used for the analysis of all statistical tests in this study. Descriptive statistics, including mean, standard deviation, and frequency were used to describe the nurses' levels of self-esteem, interpersonal relationship, sense of symbolic immortality, death anxiety, and ageism as well as sociodemographic and professional characteristics. Independent t-tests were used for comparisons between the intervention and control groups in the main variables of interest. For comparisons between the pre and posttest scores of nurses in both groups, paired t-tests were used. Hierarchical multiple regression was used to examine the significant predictors of nurses' ageism. The order of entry of the variables into the regression model was based on their order in the TMT. Death anxiety was entered in the final step into the regression model as it is the main independent variable of ageism.

ELIGIBILITY:
Inclusion Criteria:

* The eligible participants in this study were nurses caring for older adults and working in the hospital for at least one year of clinical experience.

Exclusion Criteria:

* Nurses working in Pediatric, maternity, and psychiatric departments
* Nurses with clinical experience less than one year

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Ageism | Two months
  The Fraboni Scale of Ageism (FSA) (Fraboni et al., 1990) was used to measure nurses' ageist attitudes toward older adults. The FSA is a 29-item scale measuring the attitudinal and affective aspects of ageism. The FSA has three positive items (e.g., "Old people can be very creative"), which were reverse coded before calculating the total score. Each item of the FSA has four possible responses, including: "1= strongly disagree,"; "2= disagree,"; " 3=agree,"; and " 4= strongly agree". The possible range of the total score of the FSA is from 29 to 116. Higher scores indicate greater levels of ageist attitudes. The internal consistency reliability of the FSA in this study was high (Cronbach's alpha = 0.89), which is very close to the original research (0.86) (Fraboni et al., 1990)
Death anxiety | two Months
  Death anxiety was measured using The revised Collett-Lester Fear of Death Scale (CL-FODS) (Lester & Abdel-Khalek, 2003). The CL-FODS is a 28-item scale measure death anxiety about four main aspects of death and dying, including: " your own death,"; "your own dying"; " the death of others,"; and " the dying of other". Each subscale has seven items answered on a 3-point intensity scale (ranged from 1= "no" to 5= "very"). The CL-FODS had very satisfactory reliability scores ranged from .88 to .93, and good internal consistency scores ranged from .74 to .90 in the original study. In the current study, the internal consistency reliability was satisfactory (Cronbach's alpha= 0.79)

SECONDARY OUTCOMES:
symbolic immortality | Two Months
  Symbolic immortality was measured using the Sense of Symbolic Immortality Scale (SSIS) (Drolet, 2007). The SSIS contains 11 negatives (e.g., nothing interesting happens in my life) and positive (e.g., I feel that I am doing what I want in life) items about areas of life showing the desire for symbolic immortality. The nurses responded to these items using a Likert scale of five choices ranging from 1 = "strongly disagree," to 5 = "strongly agree." The total score of the SSIS was calculated after reverse coding the negative items, yielding a range from 26 to130. Higher scores indicate a greater sense of symbolic immortality. The SSIS had good internal consistency in this study (Cronbach alpha = 0.86).
self-esteem | two Months
  Nurses' self-esteem was measured using the Rosenberg Self-Esteem Scale (RSES) (Rosenberg, 2015). The RSES has five positive (e.g., "I take a positive attitude toward myself") and five negatives (e.g., "I feel I do not have much to be proud of") items. The nurses responded to these items using a 4-point Likert scale ranging from 1= "strongly disagree" to 4= "strongly agree." The total score of the RSES was calculated after reverse coding of the negative items yielding a range from 10 to 40, with higher scores indicating greater levels of self-esteem. The Cronbach's alpha reliability of the RSES in this study was high (0.91)
interpersonal relationship | two Months
  Nurses' interpersonal relationships were measured using the Interpersonal Reactivity Index (IRI) (Davis, 1980). The IRS has four subscales consisting of five positive and two negative items each. The subscales include perspective-taking, fantasy, empathic concern, and personal distress. The nurses responded to the 28 items of IRS with five responses ranging from 0=" Does not describe me well" to 4= "describes me very well." The total score of the IRS was calculated after reverse coding the negative items, yielding a range from 0 to 112. The Cronbach's alpha reliability of the IRI in this study was very good (0.81)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Rababa, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- King Abdullah University Hospital, Irbid, Jordan

REFERENCES:
- [Derived] Rababa M, Alhawatmeh H, Al Ali N, Kassab M. Testing the Effectiveness of Cognitive Behavioral Therapy in Relieving Nurses' Ageism Toward Older Adults: A Randomized Controlled Trial. Cognit Ther Res. 2021;45(2):355-366. doi: 10.1007/s10608-020-10167-4. Epub 2020 Oct 20. PMID 33100426